CLINICAL TRIAL: NCT02712060
Title: Obstructive Sleep Apnoea in Children and Adolescents With Ehlers-Danlos Syndrome
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Children's Hospital, Zurich (Other); Ehlers-Danlos Network, Switzerland (Other)
Responsible Party: Principal Investigator, Malcolm Kohler, Prof. Dr. med., University of Zurich
Other Study IDs: KEK-ZHNr. 2015-0144
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Ehler's Danlos Syndrome; Obstructive Sleep Apnea
Keywords: Ehlers-Danlos Syndrome; Obstructive Sleep Apnea; Prevalence; Children; Pediatric; Adolescents
MeSH Terms: conditions — Sleep Apnea, Obstructive; Ehlers-Danlos Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EDS patients: Patients with the diagnosis of Ehlers-Danlos syndrome
  Interventions: Other: No intervention
- controls: Patients/Subjects without the diagnosis of Ehlers-Danlos syndrome
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Ehlers-Danlos Syndrome (EDS) is a clinically and genetically heterogeneous group of inherited connective tissue disorders characterized by joint hypermobility, skin hyperextensibility, and tissue fragility. EDS features such as genetically related cartilage defects, craniofacial abnormalities and increased pharyngeal collapsibility have been proposed to cause obstructive sleep apnoea (OSA). There is evidence from studies based on questionnaires that EDS patients might be more frequently affected by OSA and sleep disturbances than the general population. However, the actual prevalence of OSA in children and adolescents with EDS is unknown.

The primary objective of this study is to assess the prevalence of OSA in children and adolescents with EDS (25) compared to a matched control group (25). The secondary objective of this pioneer study is to assess the quality of life in children and adolescents in EDS in comparison to healthy children and adolescents.

DETAILED DESCRIPTION:
Ehlers-Danlos Syndrome (EDS) is a clinically and genetically heterogeneous group of inherited connective tissue disorders characterized by joint hypermobility, skin hyperextensibility, and tissue fragility. EDS features such as genetically related cartilage defects, craniofacial abnormalities and increased pharyngeal collapsibility have been proposed to cause obstructive sleep apnoea (OSA). There is evidence from studies based on questionnaires that EDS patients might be more frequently affected by OSA and sleep disturbances than the general population. However, the actual prevalence of OSA in children and adolescents with EDS is unknown.

The primary objective of this study is to assess the prevalence of OSA in children and adolescents with EDS compared to a matched control group. The secondary objective of this pioneer study is to assess the quality of life in children and adolescents in EDS in comparison to healthy children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Diagnosis of Ehlers-Danlos Syndrome (not for control group)

Exclusion Criteria:

* Moribund or severe disease prohibiting protocol adherence
* Continuous positive airway pressure treatment for OSA during sleep study
* Physical or intellectual impairment precluding informed consent or protocol adherence
* Pregnant patients

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Prospective case-control study including children and adolescents from 0-18 with EDS and matched controls. The following outcomes will be assessed: 1) apnoea-hypopnoea index, 2) sleep-related questionnaires, 3) medical chart review
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of OSA in children and adolescents with EDS | up to 12 months

SECONDARY OUTCOMES:
Quality of life in children and adolescents with EDS | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Principal Investigator — University of Zurich
Locations (1):
- Division of Pulmonology, University Hospital Zurich, Zurich, Switzerland